CLINICAL TRIAL: NCT03805152
Title: A 48-Week Prospective, Double-Blinded, Randomized, Cross-over Design in Multicenter Study of 250 Unit of Dysport Versus 50 Unit of Neuronox Injection For Cervical Dystonia in Thai Patients
Brief Title: Abobotulinum Toxin and Neubotulinum Toxin Injection in Cerivical Dystonia
Acronym: DNCD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Principal Investigator, Dr Subsai Kongsaengdao, Associated Professor, Department of Medical Services Ministry of Public Health of Thailand
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A-01-2019
Record Dates: First submitted 2019-01-08; First posted 2019-01-15 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Injections, Intramuscular; abobotulinumtoxinA

STUDY DESIGN:
Intervention Model Description: Double Blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Complete blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuronox(R) intramuscular injection (Active Comparator): Neu-botulinum Toxin Type A (Neuronox(R) - botulinum toxin type A product by medyceles company , Korea) 50 units Intramuscular injection in the affected neck muscle that cause cervical dystonia every 12 weeks for 24 weeks ( 2 times , 12 week interval)
  Interventions: Drug: Neuronox(R)
- Dysport (R) intramuscular injection (Active Comparator): Abo-botulinum Toxin Type A (Dysport (R) - botulinum toxin type A product by IPEN company, France ) 250 unit Intramuscular Injection in the affected neck muscle that cause cervical dystonia every 12 weeks for 24 weeks (2 times , 12 week interval)
  Interventions: Drug: Dysport (R)

INTERVENTIONS:
Drug: Neuronox(R) — Injection botulinum toxin intramuscular for affected neck muscle
  Other Names: Intramuscular injection
  Arms: Neuronox(R) intramuscular injection
Drug: Dysport (R) — Intramuscular injection
  Arms: Dysport (R) intramuscular injection

SUMMARY:
A 48-Week Prospective, Double-Blinded, Randomized, Cross-over design in Multicenter Study of, 250 unit of Abobotulinum Toxin Type A (Dysport) and 50 unit of Neubotulinum Toxin Type A (Neuronox) injection for Cervical Dystonia in patient diagnosed with cervical dystonia according to clinical diagnosis. It was designed to evaluate the efficacy, safety, tolerability, quality of life and the comparesion the improvement after treatment by of Abobotulinum Toxin Type A (Dysport) injection versus Neubotulinum Toxin Type A (Neuronox)Injection.

DETAILED DESCRIPTION:
Abobotulinum neurotoxin type A, abo-BoNT/A, (Dysport®) is the most potent biological toxin produced from Clostridium botulinum. In 1920, Dr Hermann Sommer of the Hooper Foundation at the University of California made the first attempt to purify the botulinum toxin. His work paved the way for further studies at Cam (Fort) Detrick on botulinum toxin type B, C, D, and E, particularly during the World War II. In 1946, Dr Carl Lammanna first crystalised the botulinum toxin type A and found it was composed of toxic units bound to non-toxic unit proteins. Dr Vernon Brooks, suggested that the botulinum toxin type A might be use to reduce the activity of hyperactive muscle in 1950s (9). In 1970-1971 Dr Alan B. Scott evolved an elegant electrophysiology EMG-guided technique to inject small doses of various agents to produce weakening of extraocular muscle for non-surgical treatment of strabismus. By 1973, he demonstrated in animal experiments that botulinum can be used for the treatment of strabismus and suggested that it might be of benefit for treating blepharospasm. In 1977, the U.S.FDA approved the botulinum toxin for human study and the result of the first clinical trial of botulinum toxin for strabismus was published in 1980. The U.S. FDA approved the botulinum toxin treatment in various movement disorders in 1990.

In 1991, the United Kingdom authorized the licence of Dysport®, and was commercially marketed by Speywood Pharmacuticals Ltd (previously Porton Products Ltd). After it's initial success in the treatment of strabismus, Botulinum toxin was used to treat other ophthalmological conditions, such as dysthyroid ophthalmopathy (1) and nystagmus (2) blepharospasm (3), focal abnormal movement such as hemifacial spasm, spasmodic torticollis, spasticity such as dystonia and pain such as cervical and lumbar pain (4).

There has been a steady stream of ideas for other uses, such as urinary, rectal, gastroesophageal sphincter and sphincter of Oddi disturbances, cosmetic (reduction of wrinkle) and eventually tension-type headache. In the past few years, some clinical observation from Brin, MasKop reported that patients who had been injected with botulinum toxin for wrinkle had some benefit for relieving headache. Three documented studies showed the clinical use of botulinum toxin for migraine prophylaxis.(26) Neubotulinum Toxin Type A, (Neu-BoNT/A), (Neuronox® ) (Medytox Inc, Ochang-eup, Cheongwon-gu, Cheongju-si, Chungcheongbuk-do, Republic of Korea), also known as Meditoxin in Korea, is a newly manufactured BoNT-A (Neu-BoNT/A) that was developed to provide features close to onabotulinum toxin A (5). Neuronox was tested in a murine model, and its effect on muscle force generation was equivalent to Botox® (ona-BoNT/A) (6). A previous multicenter randomized controlled trial showed that Neuronox and Botox® have equivalent efficacy and safety for the treatment of spastic equinus in children with cerebral palsy (6). However, Neuronox has not yet been investigated in post-stroke upper limb spasticity and cervical dystonia.

STUDYOBJECTIVES Primary Objective Comparesion of pre- and post- treatment after 12 and 24 week TWSTRS and CDIP-58 scale with 50 unit of Neubotulinum Toxin Type A (Neuronox) and 250 unit of Abobotulinum Toxin Type A (Dysport) incervical dystonia patients 8.2 Secondary Objective Comparesion the quality of life (SF 36, CES-D) pre- and post- 12 and 24 week treatment with 50 unit of Neubotulinum Toxin Type A (Neuronox) and 250 unit of Abobotulinum Toxin Type A (Dysport) incervical dystonia patients There were two treatment arms in crossover designed study and the interest was only on the comparison of each pre- and post- treatment outcomes of (Dysport)and (Neuronox) , two pair- wise comparisons pre and post treatment after 12 and 24 week scale were carried out. For each of the pair-wise comparison, 2-sided p-value was used to ensure that the overall Type I error=0.05. Beta error 80% Multiple repeated analysis and general linear model will be analysed in the efficacy of treatment.Two-sided exact p-values were reported in the efficacy analyses. Demographic and safety analyses were based on the summary of descriptive statistics.

At the screening visit and prior to performance of any study procedures, the investigators would explain the details of the study and the subject would have to sign on the written informed consent, exclusion criteria, and inclusion criteria Each subject who was willing to enrol into the study was asked about their medical history as well as their recent and current medications being taken.

All enrolled subjects were asked to undertake an initial physical examination and had to satisfy the criteria for the inclusion /exclusion before being enrolled into the study.

All patients were asked to complete physical examination, TWSTRS, CDIP-58, SF36, PHQ9 and CES-D .

Laboratory blood (livers tests, haematology,) examinations, urine pregnancy test) were performed for safety reasons.

1Inclusion Criteria The subjects need to satisfy the following criteria before being allowed to participate in the study:

* The subject has to grant permission to enter into the study by signing and dating the informed consent form before completing any study-related procedure such as any assessment or evaluation not related to the normal medical care of the subject.
* Able to give written inform consent and retained one copy of the consent form • Male or female subject, aged between 18 - 100 years old.
* Subject diagnosed to be cervical dystonia.
* Female subject in good health and sexually active was instructed by the investigator to avoid pregnancy during the study and to use condom or other contraceptive measure if necessary. The subject was required to have a negative urine pregnancy test before being eligible for the study. (At each of the subsequent visit, a urine pregnancy test was performed).
* Subject judged to be reliable for compliance for taking medication and capable of recording the effects of the medication and motivated in receiving benefits from the treatment.

Subject should undergo a normal physical and neurological examination TWSTRS, CDIP-58, SF36, and CES-D

* during the whole study period at will. 9.2.2 Exclusion Criteria The subject WERE NOT ALLOWED TO enter/continue into the study, if :.
* The subject was pregnant or lactating.
* The subject was a female at risk of pregnancy during the study and not taking adequate precautions against pregnancy.
* The subject had a known hypersensitivity to any of the test materials or related compounds.
* The subject was unable or unwilling to comply fully with the protocol.
* The subject received any unlicensed drug within the previous 6 months.
* Treatment with investigational drug (s) within 6 months before the screening visit. • The subject had previously entered in this study.
* Subject with past history of botulism, other neuromuscular disorder (e.g. myasthenia gravis, Lambert - Elton Syndrome)
* Subject with significant medical / neurological / psychiatric disorders such as blood dyscrasia, thrombocytopenia, rheumatoid arthritis, congestive heart failure, coronary artery heart diseases, dementia, psychosis, or other conditions which could influence the clinical trial.
* Known history of drug abuse (narcotic (s), cafergot, or others) or drug (botulinum toxin type A) allergy.
* Unable to cooperate fill-up TWSTRS, CDIP-58, SF36, and CES-D • Patient who planned to schedule elective surgery during the study.
* The used of aminoglycoside antibiotics and curare were not allowed during the study.

ELIGIBILITY:
Inclusion Criteria:

* The subjects need to satisfy the following criteria before being allowed to participate in the study:

  * The subject has to grant permission to enter into the study by signing and dating the informed consent form before completing any study-related procedure such as any assessment or evaluation not related to the normal medical care of the subject.
  * Able to give written inform consent and retained one copy of the consent form • Male or female subject, aged between 18 - 100 years old.
  * Subject diagnosed to be cervical dystonia.
  * Female subject in good health and sexually active was instructed by the investigator to avoid pregnancy during the study and to use condom or other contraceptive measure if necessary. The subject was required to have a negative urine pregnancy test before being eligible for the study. (At each of the subsequent visit, a urine pregnancy test was performed).
  * Subject judged to be reliable for compliance for taking medication and capable of recording the effects of the medication and motivated in receiving benefits from the treatment.

Subject should undergo a normal physical and neurological examination TWSTRS, CDIP-58, SF36, and CES-D • during the whole study period

Exclusion Criteria:

- The subject WERE NOT ALLOWED TO enter/continue into the study, if :.

* The subject was pregnant or lactating.
* The subject was a female at risk of pregnancy during the study and not taking adequate precautions against pregnancy.
* The subject had a known hypersensitivity to any of the test materials or related compounds.
* The subject was unable or unwilling to comply fully with the protocol.
* The subject received any unlicensed drug within the previous 6 months.
* Treatment with investigational drug (s) within 6 months before the screening visit. • The subject had previously entered in this study.
* Subject with past history of botulism, other neuromuscular disorder (e.g. myasthenia gravis, Lambert - Elton Syndrome)
* Subject with significant medical / neurological / psychiatric disorders such as blood dyscrasia, thrombocytopenia, rheumatoid arthritis, congestive heart failure, coronary artery heart diseases, dementia, psychosis, or other conditions which could influence the clinical trial.
* Known history of drug abuse (narcotic (s), cafergot, or others) or drug (botulinum toxin type A) allergy.
* Unable to cooperate fill-up TWSTRS, CDIP-58, SF36, and CES-D • Patient who planned to schedule elective surgery during the study.
* The used of aminoglycoside antibiotics and curare were not allowed during the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Toronto Western Spasmodic Torticollis Rating scale ( TWSTRS) | 24 week
  TWSTRS ranged( 0-85 by summation of all 3 sub- scales ) higher represent a worse outcome TWSTRS Sub- scale includes
  1. TWSTRS-Total severity scale ( maximum 35 points)
  2. TWSTS-Disability scale (maximum 30 points)
  3. TWSTS-Pain scale (maximum 20 points)
Cervical Dystonia Impact Profile 58 ( CDIP-58) | 24 week
  ) Cervical Dystonia Impact Profile-58 items composed of 8 sub-scale Total score by summation of 8 subscale higher represent a worse outcome Analysis both total score (range 58-290 points) And sub-scale analysis composed of Head and neck symptoms ( 6 items ; 6-30 points) Pain and discomfort ( 5 items ; 5-25 points) Upper limb activity ( 9 items ; 9-45 points) Walking ( 9 items ; 9-45 points) Sleep ( 4 items ; 4-20 points) Annoyance ( 8 items ; 8-40 points) Mood (7 items ; 7-35 points) Psychosocial functioning ( 10 items ; 10-50 points)

SECONDARY OUTCOMES:
Comparesion the quality of life 36 item ( SF 36) | 24 week
  Comparesion the quality of life (SF 36) pre- and post- 12 and 24 week ttreatment with 50 unit of Neubotulinum Toxin Type A (Neuronox) and 250 unit of Abobotulinum Toxin Type A (Dysport) this score has special formula calculation
Depression scale measured by Center of Epidemiologic Study of Depression 20 item ( CES-D 20) | 24 week
  Comparesion of CES-D pre- and post- 12 and 24 week treatment with 50 unit of Neubotulinum Toxin Type A (Neuronox) and 250 unit of Abobotulinum Toxin Type A (Dysport) Score ranged from 20-80 points higher represent a worse outcome
Depression scale measured by Patient Health Questionnaire Depression Scale (PHQ-9) | 24 week
  Comparesion of PHQ-9 pre- and post- 12 and 24 week treatment with 50 unit of Neubotulinum Toxin Type A (Neuronox) and 250 unit of Abobotulinum Toxin Type A (Dysport) There is the special scale calculation for diagnosis Major depressive disorder, Other depressive disorder and others,higher points /score represent a worse outcome ranged 0-27 points plus 3 points Total summation of 5-9 points indicate Minimal symptoms, 10-14 Minor depression ++ or Dysthymia* or Major depression, mild , 15-19 points Major depression, moderately severe
  ≥ 20 Major depression, severe
Clinical Global Impression of Changed ( CGIC) | 24 week the scale compose of -3 to 3 higher represent a good outcome
  Comparesion of CGIC pre- and post- 12 and 24 week treatment with 50 unit of Neubotulinum Toxin Type A (Neuronox) and 250 unit of Abobotulinum Toxin Type A (Dysport)

CONTACTS AND LOCATIONS:
Overall Officials: Subsai Kongsaengdao, Principal Investigator — Division of Neurology, Department of Medicine, Rajavithi Hospital, Department of Medical services, Public Health Ministry, Bangkok, 10400 Thailand 3 Department of Medicine, College of Medicine, Rangsit University, Bangkok, 10400 Thailand
Locations (4):
- Thailand (4):
  - Assistant Professor Subsai Kongsaengdao, Bangkok
  - Lampang Hospital, Lampang
  - Surat Thani hospital, Surat Thani
  - Sappasithiprasong Hospital, Ubon Ratchathani

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kongsaengdao S, Maneeton B, Maneeton N. Quality of life in cervical dystonia after treatment with botulinum toxin A: a 24-week prospective study. Neuropsychiatr Dis Treat. 2017 Jan 10;13:127-132. doi: 10.2147/NDT.S116325. eCollection 2017. PMID 28138245
- [Background] Kongsaengdao S, Maneeton N, Maneeton B. Long-term quality of life in cervical dystonia after treatment with abobotulinum toxin A: a 2-year prospective study. Neuropsychiatr Dis Treat. 2018 Apr 26;14:1119-1124. doi: 10.2147/NDT.S152252. eCollection 2018. PMID 29731634